CLINICAL TRIAL: NCT06583421
Title: Children With High Genetic Susceptibility Benefit More From Short-term Physical Activity Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Haonan Zhou, Master student, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ethics Approval No. [2020] 075
Record Dates: First submitted 2024-08-22; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Physical Inactivity; Obesity, Childhood
Keywords: Obesity; Physical activity; Genetic susceptibility; Interaction
MeSH Terms: conditions — Sedentary Behavior; Pediatric Obesity; Obesity; Motor Activity; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-week MVPA intervention group (Experimental): The 4-week MVPA intervention engaged in supervised aerobic exercise, resistance training and interesting sport for 60 minutes, 3 days/week (Monday, Wednesday and Friday). As shown in Table S1, participants completed four sessions including preparation module (15 min), training module (30 min), and relaxation module (15 min). Another aerobic module (15 min) was added in each Friday. Children in intervention group were also encouraged to take exercise for 10 minutes together with their parents at home two hours later after dinner including ten minutes' walking (at least 1000 meters) or at least 200 times rope skipping.
  Interventions: Behavioral: 4-week MVPA intervention
- Control group (No Intervention): No physical activity interventions were conducted in the control group. In order to safeguard the rights of the control groups, the same physical activity intervention was given to the control group at the end of the research.

INTERVENTIONS:
Behavioral: 4-week MVPA intervention — The 4-week MVPA intervention engaged in supervised aerobic exercise, resistance training and interesting sport for 60 minutes, 3 days/week (Monday, Wednesday and Friday). As shown in Table S1, participants completed four sessions including preparation module (15 min), training module (30 min), and relaxation module (15 min). Another aerobic module (15 min) was added in each Friday.
  Arms: 4-week MVPA intervention group

SUMMARY:
Sharp increase in childhood obesity has been regarded as one of the most serious but preventable global public health challenges. Engaging children in moderate-to-vigorous physical activity (MVPA) is important to address the obesity problem as it is associated with a host of obesity outcomes including body weight, BMI, body fat percentage, waist circumference, lean body mass, systolic blood pressure, insulin sensitivity, cardiovascular health, and cognitive development. In China, only about one-third of children meet the recommended guidelines of at least 60 minutes of MVPA per day, and obesity rates are rising.

Children with different generic characteristics may benefit differently from MVPA, which should not be neglected when conducting interventions among children. However, most of the evidence about how genes interact with MVPA on obesity among children were addressed from cross-sectional design or synthetic lifestyle interventions. Change-on-change analysis was used in our study based on a randomized controlled trial of MVPA intervention to discusses the effect of genetics and physical activity on obesity indicators. In addition, investigators used Generic risk scores (GRSs) based on 14 BMI-associated SNPs to assess generic variation of Chinese children.

DETAILED DESCRIPTION:
This study is based on a randomized controlled trial of a 4-week MVPA intervention. PASS 11.0 software was used to calculate the sample size of the randomized controlled trial study (quantitative variable). Investigators recruited obese children aged 10-12 years according to the criteria for overweight and obesity in Chinese children and adolescents proposed by the Working Group on Obesity in China (WGOC). Children with physical activity-limiting diseases and obesity due to diseases were excluded.

The 4-week MVPA intervention engaged in supervised aerobic exercise, resistance training and interesting sport for 60 minutes, 3 days/week (Monday, Wednesday and Friday). No physical activity interventions were conducted in the control group. In order to safeguard the rights of the control groups, the same physical activity intervention was given to the control group at the end of the research.

Physical activity strength was measured by Tri-axial body motion recorder (ActiGraph, Wgt3x-BT, USA) to maintain relative intensity. At baseline, Physical Activity Questionnaire for Children (PAQ-C) was answered by each participant.

Height was measured to the nearest 0.1cm using Height Measuring Ruler (Selcom, Germany). Body weight and fat mass was measured to the nearest 0.1kg using Body Composition Analyzer (DC-13, Parade, Japan).Waist circumference and hip circumferencewas measured to the nearest 0.1cm with measuring tape.

Preperitoneal fat and abdominal subcutaneous fat thickness were measured by ultrasonography. The thickness and area of preperitoneal fat and abdominal subcutaneous fat were measured with a linear array probe L12-5 (38 mm, 5-12 HZ) according to the method of Suzuki.

The whole genomic DNA of blood mononuclear cells was performed using a fully automated nucleic acid extractor (QIAGEN, QIAcube, Germany), the DNA extraction reagents were used in a magnetic bead method DNA extraction kit (QIAGEN, 51331, Germany), and the detailed steps were performed according to the reagent and instrument instructions. 14 SNP loci associated with obesity and BMI were reliably validated based on GWAS studies in large Asian populations.

ELIGIBILITY:
Inclusion Criteria:

* obese children aged 10-12 years

Exclusion Criteria:

* obesity due to disease
* persons with limited physical activity

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Physical activity strength | During the 4-week intervention
  Strength was measured by Tri-axial body motion recorder (ActiGraph, Wgt3x-BT, USA) to maintain relative intensity. Children were required to wear ActiGraph by a professional investigator on the left wrist, loosely tightened, and required to wear it at all times except for the shower during the intervention for 7 days.
Height | At baseline and after 4-week of intervention
  eight was measured to the nearest 0.1cm using Height Measuring Ruler (Selcom, Germany).
Body weight | At baseline and after 4-week of intervention
  Body weight was measured to the nearest 0.1kg using Body Composition Analyzer (DC-13, Parade, Japan)
Fat mass | At baseline and after 4-week of intervention
  Fat mass was measured to the nearest 0.1kg using Body Composition Analyzer (DC-13, Parade, Japan).
Waist circumference | At baseline and after 4-week of intervention
  Waist circumference was measured to the nearest 0.1cm with measuring tape.
Hip circumference | At baseline and after 4-week of intervention
  Hip circumference was measured to the nearest 0.1cm with measuring tape.
Preperitoneal fat | At baseline and after 4-week of intervention
  Preperitoneal fat was measured by ultrasonography. The thickness and area of preperitoneal fat was measured with a linear array probe L12-5 (38 mm, 5-12 HZ) according to the method of Suzuki.
Abdominal subcutaneous fat thickness | At baseline and after 4-week of intervention
  Abdominal subcutaneous fat thickness was measured by ultrasonography. The thickness and area of abdominal subcutaneous fat was measured with a linear array probe L12-5 (38 mm, 5-12 HZ) according to the method of Suzuki.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Shenyang, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT06583421/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT06583421/ICF_001.pdf